CLINICAL TRIAL: NCT06026397
Title: A Randomized, Double-blind, Placebo-controlled, Sequential Dose-escalation Clinical Study to Evaluate the Safety and Tolerability of SK10 Powders (Inactivated Bacteroides Fragilis) in Healthy Adult Subjects
Brief Title: A Sequential Single and Multiple Ascending Dose (SAD/MAD) Study of SK10 Powders in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Zhiyi Biotechnology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SK10-101
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Chemotherapy-induced Diarrhea
Keywords: Single ascending dose; Multiple ascending dose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants will receive dose A of SK10 (n=6) or placebo (n=2)
  Interventions: Drug: SK10; Drug: Placebo
- Cohort 2 (Experimental): Participants will receive dose B of SK10 (n=6) or placebo (n=2)
  Interventions: Drug: SK10; Drug: Placebo
- Cohort 3 (Experimental): Participants will receive dose C of SK10 (n=6) or placebo (n=2)
  Interventions: Drug: SK10; Drug: Placebo

INTERVENTIONS:
Drug: SK10 — Participants will be randomized to receive oral suspension of SK10 powder, includes SAD on Day 1 and 14-days MAD from Day 4 to Day 17.
Drug: Placebo — Participants will be randomized to receive oral suspension of placebo, includes SAD on Day 1 and 14-days MAD from Day 4 to Day 17.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of orally administered SK10 powders in healthy adult subjects at three dose levels, following single and multiple doses.

DETAILED DESCRIPTION:
This is a first-in-human, Phase 1, randomized, double-blind, placebo-controlled, sequential SAD and MAD study to assess the safety and tolerability of orally administered SK10 powders in healthy adult subjects.

This is a dose escalation study with three sequential cohorts planned testing at 3 dose levels.

A total of 24 subjects are planned to be enrolled into 3 cohorts (Cohorts 1, 2 and 3). Within each cohort, eligible subjects will be randomized to receive SK10 or placebo in a 3:1 ratio. The treatment duration includes a single dose administration on Day 1 and 14-day repeat doses administration from Day 4 to Day 17.

The study consists of:

* Screening Period (28 days [Day -28 to Day -1])
* Treatment Period (Day -1 to Day 19)
* Follow-up Visit (Day 24).

The study duration will be approximately up to 52 days, conducted at a single center.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have negative test results for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), anti-hepatitis C virus antibodies (anti-HCV) and anti-human immunodeficiency virus (HIV) antibodies at Screening Visit
* Body weight ≥ 50.0 kg for males, or ≥ 45.0 kg for females, and body mass index within the range of 18.0-28.0 kg/m2 (inclusive).
* A male subject must agree to use together with his female partner/ spouse a highly effective contraception form of birth control in combination with a barrier method throughout the clinical study period and until 90 days after the last dose of IMP. Male subjects must also refrain from donating sperm from the time of informed consent until 90 days after the last dose of IMP.
* A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Non-childbearing potential (OR)
  * A woman of childbearing potential (WOCBP) who agrees to use highly effective methods of birth control in combination with a barrier method at least 3 months prior to the Screening Visit until 30 days after the last dose of IMP.
  * WOCBP must agree not to donate ova from the time of informed consent until 30 days after the last dose of IMP.
  * WOCBP must have a negative serum pregnancy test at the Screening Visit.

Exclusion Criteria:

* History or presence of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* History/current symptom related to gastrointestinal abnormalities within 2 weeks before the first dose.
* Subject is a pregnant or lactating women.
* Known or suspected hypersensitivity to the IMP or excipients of the IMP.
* Subjects with lactose intolerance/allergy.
* Known or ongoing psychiatric disorders, or active neuropsychiatric disease deemed clinically significant in the opinion of the investigator.
* Subject has used over-the-counter or other oral medications (including vitamins), prescription medications, or herbal remedies within 14 days before dosing.
* Subject has had major surgery within 3 months before Screening, or plan to perform surgery during the study.
* Subject experiences an acute medical condition or uses concomitant medication during the Screening period.
* Subject has been treated with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of the IMP.
* Subject has taken probiotic foods and/or drinks and/or health products within 1 week before the first dose.
* History of alcohol and/or illicit drug abuse within 2 years before Screening.
* Subject has positive urine drug or alcohol test at the Screening Visit or Admission.
* No more than 5 cigarettes are allowed from screening to admission, and smoking is not allowed from admission until after the last follow-up visit.
* Subject has donated or lost ≥ 400 mL of whole blood within 3 months or donated plasma within 14 days before Screening.
* Subjects has received vaccination within 14 days before the first dose or vaccination planned during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-11 (Actual); Study Completion 2024-02-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment-Emergent Adverse Events (TEAEs) | From screening (Day -28) up to follow-up [FU] (Days 24±2)
  Number of participants with TEAEs to evaluate the safety and tolerability of SK10 in healthy adult subjects
Number of participants with clinically relevant changes from baseline electrocardiogram (ECG) parameters | From screening (Day -28), Days -1,1,3, 11,19 up to FU (Days 24±2)
  Number of participants with clinically relevant changes from baseline ECG parameters to evaluate the safety and tolerability of SK10 in healthy adult subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Early Phase Clinical Unit (EPCU) - PAREXEL, Glendale, California, United States